CLINICAL TRIAL: NCT03633903
Title: Mindfulness for Resilience in Early Life
Acronym: MindREaL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIBR # 2018-003-00
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Adolescent With Early Life Stress; Resilience
Keywords: Early life stress; Adolescent; Mindfulness; Neurobiological; Stress; Resilience
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Adolescents are randomly assigned to either a mindfulness intervention or no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Active Comparator): Mindfulness: Eight sessions, twice per week over four weeks. Surveys administered prior to each session.
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): Treatment as usual (i.e., pharmacotherapy, psychotherapy, etc.) for the four week duration with twice weekly surveys administered.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness based stress reduction adapted for teens is a mindfulness intervention designed to aid adolescents in understanding stress, better coping with stress, and promoting resilience
  Arms: Mindfulness

SUMMARY:
Early life stress (ELS) is associated with a number of psychiatric and medical conditions later in life, thought to be caused by subsequent disruptions in biological processes involved in regulation of stress responses. Given that these alterations have long-lasting effects, there is a great need for effective preventative interventions. The long-term goal of this project is to identify early interventions that may most powerfully mitigate risk for psychiatric illness among adolescents with exposure to early life stress (ELS), with a focus on interventions that can be widely and effectively implemented, have the potential for long-lasting benefits, and can effectively engage targeted neurobiological processes and networks. The specific aims of the present study are to 1) examine how ELS impacts biological processes associated with regulation of stress, and 2) identify how MBI impacts affective symptoms and biological processes dysregulated by ELS.

This study supports the efforts to reduce the effects of early adversity in children by testing an impact of an effective psychological intervention on disrupted biological processes caused by early adversity. Successful achievement of the proposed aims will contribute to a) the knowledge base needed to reduce the effects of trauma and stress in children and families and b) the development of easily implemented and disseminated preventative interventions.

The proposed study will utilize a multi-method design to examine the effect of mindfulness on biological processes (i.e., stress responses) disrupted by exposure to ELS among adolescents age 13 to 15. Adolescents will first complete self-report measures of childhood adverse experiences, trauma, and neglect. Forty eligible adolescents will be next randomly assigned to either an eight session mindfulness-based stress reduction intervention for teens or no treatment. Pre- and post-intervention assessment will include (a) self-report measures of symptoms and emotion regulation, (b) a blood draw for assessment of inflammatory markers and gene expression, and (c) a stress task with saliva cortisol collected before and after this task.

ELIGIBILITY:
Inclusion Criteria:

* Age 13.00 to 15.99 years at time of baseline assessment
* Able to validly and safely complete baseline assessments
* All genders
* All races
* Eligibility as a subject with early life stress will be determined by:
* Scoring 4 or greater on Adverse Childhood Experiences (ACE) scale, with at least two experiences having occurred prior to age 10.

Exclusion Criteria:

* No biological parent or legal guardian identified to give permission for minor to participate
* History of neurological disorders including seizure disorder, cerebral palsy, or other conditions requiring neurological or medical care, being managed for migraines (e.g., daily prophylactic medication, seeing a neurologist for migraines), or a diagnosis of Developmental Delay, including severe learning disorder, mental retardation, pervasive developmental disorder, or other conditions requiring repeated and persistent specialized education.
* Current psychotic disorder, bipolar disorder, obsessive-compulsive and related disorders, substance use disorder, or conduct disorder.
* Current active suicidal ideation.
* Current use of medications with major effects on brain function or blood flow (e.g., antipsychotics, mood stabilizers); ADHD medications and SSRIs, that have been stable for at least 6 weeks, are not exclusionary since their use is associated with conditions that confer risk for monitored disorders that emerge in adolescence, and assessment of these individuals will provide useful data to the scientific community. Youth on ADHD medications and SSRIs will not be asked to go off their medications.
* Not fluent in English
* Non-correctable vision, hearing or sensorimotor impairments, as protocol elements may not be valid.
* Youth planning to move to an area not within reasonable traveling distance of LIBR; knowledge at baseline that treatment completion / follow-up will not be possible.
* Youth appears to be high/intoxicated, or withdrawing from the effects of alcohol or drugs at time of enrollment.
* Youth / parent who are unable or unwilling to provide biological samples (i.e., blood draws or saliva collection).
* Female youth who are pregnant
* Youth who are currently in unsafe environments (e.g., currently living with an abusive parent)

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namik Kirlic, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen ZP, Cosgrove KT, Akeman E, Coffey S, Teague K, Hays-Grudo J, Paulus MP, Aupperle RL, Kirlic N. The effect of a mindfulness-based stress intervention on neurobiological and symptom measures in adolescents with early life stress: a randomized feasibility study. BMC Complement Med Ther. 2021 Apr 15;21(1):123. doi: 10.1186/s12906-021-03295-1. PMID 33858395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents and their families were recruited from the community using flyers, radio advertisements, billboards, and a school-based messaging platform (e.g., PeachJar).
Groups:
- Mindfulness: Mindfulness: Eight sessions, twice per week over four weeks
  Mindfulness: Mindfulness based stress reduction adapted for teens is a mindfulness intervention designed to aid adolescents in understanding stress, better coping with stress, and promoting resilience
- Control: Treatment as usual, inactive control group
Period: Overall Study
Arm/Group | Mindfulness | Control
Started | 22 | 18
Intent to Treat | 0 | 18
Completed | 16 | 11
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Control | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two subjects were removed from analyses due to not beginning intervention or control group.
  years
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 14.33 (0.73) | 14.29 (0.77) | 14.31 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two subjects were removed from analyses due to not beginning intervention or control group.
  Participants
    number analyzed (Participants) | 21 | 17 | 38
    Female | 7 | 8 | 15
    Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two subjects were removed from analyses due to not beginning intervention or control group.
  Participants
    number analyzed (Participants) | 21 | 17 | 38
    Hispanic or Latino | 2 | 1 | 3
    Not Hispanic or Latino | 19 | 16 | 35
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two subjects were removed from analyses due to not beginning intervention or control group.
  Participants
    number analyzed (Participants) | 21 | 17 | 38
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 5 | 9
    White | 10 | 9 | 19
    More than one race | 5 | 0 | 5
    Unknown or Not Reported | 0 | 1 | 1
Change in salivary cortisol [Mean (Standard Deviation); unit: μg/dL] — This measure is the change in cortisol from the stress induction task. Salivary cortisol was collected 20 minutes before and 20 minutes after stress induction. For analyses, we subtracted post minus pre cortisol levels, such that negative values are possible if post stress induction cortisol was lower than pre stress induction cortisol. Population: Two subjects were removed from analysis due to not beginning intervention or control.
  μg/dL
    baseline, pre stress induction: number analyzed (Participants) | 21 | 17 | 38
    baseline, pre stress induction | 0.12 (0.89) | -0.16 (1.15) | -0.02 (1.02)
    baseline, post stress induction: number analyzed (Participants) | 21 | 17 | 38
    baseline, post stress induction | -0.22 (0.88) | 0.27 (1.10) | 0.025 (0.99)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — Population: Two subjects were removed from analysis due to not beginning intervention or control.
  mg/L
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 1.16 (3.82) | 2.39 (5.75) | 1.775 (4.785)
Interleukin-6 [Mean (Standard Deviation); unit: pg/mL] — Population: Two subjects were removed from analysis due to not beginning intervention or control.
  pg/mL
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 0.47 (0.48) | 0.83 (1.19) | 0.65 (0.835)
Depression and Anxiety Symptoms [Mean (Standard Deviation); unit: units on a scale] — We used the Mood and Feelings Questionnaire - Short Form (MFQ-sf) to characterize symptoms of anxiety and depression. The MFQ-sf is a 13-item questionnaire with a simple sum score for the entire scale. Minimum score = 0, maximum score = 26. Scores of 8 or more indicate moderate depression.
  Codings reflect whether the phrase was descriptive of the subject most of the time, sometimes, or not at all. Higher scores indicate greater symptoms of anxiety/depression, while lower scores indicate less anxiety/depression. Population: Two subjects were removed from analysis due to not beginning intervention or control.
  units on a scale
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 6.81 (4.53) | 9.39 (6.54) | 8.1 (5.53)

OUTCOME MEASURES:

1. Primary Outcome: Cortisol Reactivity
Description: Change in level of cortisol in saliva following a social stress test. Subjects completed the Trier Social Stress Test for Children (TSST-C) at baseline and follow-up. The TSST-C consists of public speaking and serial subtraction components in front of two research confederates. The test takes approximately 20 minutes to complete. Salivary cortisol was collected 20 minutes prior to TSST-C, and 20 minutes following the end of the TSST-C, such that the TSST-C task with data collection spanned approximately one hour.
Time Frame: Baseline (pre-intervention); Follow-up (post-intervention) at 6-8 weeks from baseline
Population: Two subjects were removed from all analyses due to not having usable baseline data and withdrawing prior to intervention. One was removed from each group, such than N=22-1=21 analyzed for mindfulness and N=18-1=17 for control.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Mindfulness | Control
Number analyzed (Participants) | 21 | 17
μg/dL
  follow-up, pre stress induction | -0.21 (1.05) | 0.34 (0.85)
  follow-up, post stress induction | 0.05 (1.16) | -0.08 (0.76)
Statistical Analysis 1: Comparison: Mindfulness vs Control; Test type: Superiority; p < .05, Mixed Models Analysis — The reported p-value was calculated and is not indicating a threshold for significance. This applies to the change from row 1 to row 3 (e.g., baseline pre TSST-C versus follow-up timepoint pre TSST-C); Mean Difference (Final Values) = 1.04
Statistical Analysis 2: Comparison: Mindfulness vs Control; Test type: Superiority; p < .05, Mixed Models Analysis — The reported p-value was calculated and is not indicating a threshold for significance. This is for the difference from row 1 to row 2 (baseline pre versus baseline post TSST-C); Mean Difference (Final Values) = 0.77
Statistical Analysis 3: Comparison: Mindfulness vs Control; Test type: Superiority; p = 0.40, Mixed Models Analysis — The reported p-value was calculated and is not indicating a threshold for significance. Comparing row 1 and row 4 (baseline pre TSST-C versus follow-up post TSST-C); Mean Difference (Final Values) = 0.38

2. Primary Outcome: Immune System Activity
Description: Change in level of interleukin 6 (IL-6) and C-reactive protein (CRP) in blood
Time Frame: Baseline (pre-intervention); Follow-up (post-intervention) at 6-8 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL; mg/L
Arm/Group | Mindfulness | Control
Number analyzed (Participants) | 21 | 17
pg/mL; mg/L
  CRP (followup) | 0.83 (1.45) | 0.99 (1.32)
  I'll-6 (followup) | 0.46 (0.32) | 0.66 (0.65)
Statistical Analysis 1: Comparison: Mindfulness vs Control; Comparing group differences (CRP biomarker) in mindfulness versus control at baseline versus follow-up timepoints; Test type: Superiority; p = .39, Mixed Models Analysis; Mean Difference (Final Values) = -0.35
Statistical Analysis 2: Comparison: Mindfulness vs Control; Comparing group differences (IL-6 biomarker) in mindfulness versus control at baseline versus follow-up timepoints; Test type: Superiority; p = .95, Mixed Models Analysis; Mean Difference (Final Values) = -0.02

3. Secondary Outcome: Mood and Feelings Questionnaire
Description: Measure Description: We used the Mood and Feelings Questionnaire - Short Form (MFQ-sf) to characterize symptoms of anxiety and depression. The MFQ-sf is a 13-item questionnaire with a simple sum score for the entire scale. Minimum score = 0, maximum score = 26. Scores of 8 or more indicate moderate depression.
  Codings reflect whether the phrase was descriptive of the subject most of the time, sometimes, or not at all. Higher scores indicate greater symptoms of anxiety/depression, while lower scores indicate less anxiety/depression.
Time Frame: Baseline (pre-intervention); Follow-up (post-intervention) at 6-8 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness | Control
Number analyzed (Participants) | 21 | 17
units on a scale | 3.82 (4.61) | 8.17 (8.07)
Statistical Analysis 1: Comparison: Mindfulness vs Control; Comparing group differences (symptoms of anxiety/depression) in mindfulness versus control at baseline versus follow-up timepoints; Test type: Superiority; p = .08, Mixed Models Analysis — the calculated p value; Mean Difference (Final Values) = 0.13

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout baseline (T1), 8 sessions of twice-weekly intervention where survey responses were recorded and the MBSR-T group had group intervention (T2-T9), and follow-up (T10).
Description: No adverse events were reported or observed.
Arm/Group | Mindfulness | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03633903/Prot_SAP_000.pdf